CLINICAL TRIAL: NCT07011355
Title: The Effect of Stress Ball Use on Labor Pain and Birth Experience in Primiparous Women in the During Labor; Randomized Controlled Trial
Brief Title: Effect of Stress Ball Use on Labor Pain and Birth Experience in Primiparous Women During Labor
Acronym: stressball
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Collaborators: Sanliurfa Harran University (Unknown)
Responsible Party: Principal Investigator, Sibel Kucuk, öğretim görevlisi, Harran University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Harran-sbl-44
Record Dates: First submitted 2025-05-15; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Examine the Effect of Stress Ball Use During the Intrapartum Period on Labor Pain and Childbirth Experience in Primiparous Women
Keywords: stress ball; Primiparous; Intrapartum; Labor pain; Birth experience
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: The data will be collected after the informed consent form is signed by the women who meet the study criteria and agree to participate, after explaining the purpose of the study and the method application. The stress ball used in the study should be placed in the palm of the hand, approximately 6 cm in diameter, round, medium hardness and made of high quality silicone. While explaining the method application and its purpose, women will be addressed as squeeze ball in order to avoid negative connotations. A sufficient number of stress balls will be provided by the researchers and given to the women. During each contraction, the woman will be asked to squeeze the ball in her palm for about 3-4 seconds and then relax her hands for about 3-4 seconds. She will be asked to take a deep breath every time she squeezes the ball and exhale during relaxation. She will be asked to rest her hands between contractions (during the resting phase).
Who Masked: Outcomes Assessor
Masking Description: To avoid bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Stress ball application is an effective and non-pharmacological pain management method used during labour. Pregnant women in the intervention group are given a sterile stress ball during the active phase of labour (when the cervical opening is 1-4 cm ve 5-7 cm) and asked to squeeze this ball during uterine contractions. The main aim of this intervention is to distract the woman from pain, promote relaxation and reduce pain perception through sensory-motor stimulation.
  The stress ball squeezing movement activates the parasympathetic nervous system by interacting with the nervous system through proprioceptive sensations; this contributes to decreased muscle tone, reduced stress and relaxation. In addition, thanks to this practice, the woman's active participation in birth is supported, her perception of control over her own body increases and the birth experience is perceived more positively.
  Interventions: Other: Stress Ball
- Control group (No Intervention): Women in the will not be subjected to any practice other than routine hospital practices. The pain of each woman will be assessed and recorded by a midwife independent of the study using VAS (VAS assessment will be performed before and after contractions in the phases occurring in the first stage of labour). Data collection form The same forms will be used as for the intervention group

INTERVENTIONS:
Other: Stress Ball — Targeted Sensory Stimulus Type - Proprioceptive Input Based Mechanism:
  Stress ball application is aimed at regulating the nervous system, especially through proprioceptive and tactile (tactile) stimuli. In this respect, it differs from methods such as aromatherapy, music therapy or breathing exercises, which are more effective through the sensory, emotional or autonomic nervous system.
  Arms: Intervention group

SUMMARY:
INTRODUCTION Childbirth is a significant life experience for women, both physiologically and psychologically. The pain experienced during labor can vary depending on individual differences, cultural factors, and the course of labor. Labor pain may lead to fear, anxiety, and negative birth experiences in many women (Lowe, 2002). Therefore, using effective and safe methods to reduce pain during labor supports both maternal and fetal health and contributes to a more positive birth experience.

In recent years, non-pharmacological methods have been reported to be effective in reducing labor pain. These include breathing exercises, relaxation techniques, massage, aromatherapy, hot-cold applications, and tactile stimuli (Smith et al., 2018). The use of a stress ball is also considered one of these techniques. This method, which involves squeezing and releasing the hand, aims to promote muscle relaxation, reduce pain, and help individuals cope with stress.

This study aims to evaluate the effect of stress ball use during the active phase of labor on labor pain and the childbirth experience among primiparous women. The findings obtained may contribute to the literature by demonstrating the effectiveness of stress balls as a non-invasive intervention that can be implemented by nurses and midwives during labor.

MATERIAL AND METHODS Study Design This research is designed as a randomized controlled experimental study. It will be conducted between September and December 2025 with primiparous women admitted to the delivery unit of a public hospital in Turkey.

Population and Sample The study population will consist of primiparous women in the active stage of labor. A simple random sampling method will be used, and 64 primiparous women who meet the inclusion criteria and agree to participate in the study will be included. Participants will be randomly assigned to the intervention group (n=32) or the control group (n=32).

Ethical Approval and Informed Consent The study will be conducted after receiving approval from the [University/Hospital] Ethics Committee (Approval No: ...). Written permission to use the Childbirth Experience Questionnaire (CEQ) will be obtained from the scale's developer via email. After informing the participants about the study, those who meet the inclusion criteria and agree to participate will be asked to sign an "Informed Consent Form." The research will be carried out in accordance with the principles of the Declaration of Helsinki.

DATA COLLECTION PROCESS Data collection will begin in the latent phase of labor (cervical dilation 1-4 cm). In each phase (active phase, transition phase), participants will be instructed to squeeze the stress ball during contractions accompanied by deep inhalation and to release it during exhalation. During non-contraction periods, their hands will be rested. Participants in the intervention group will be given brief training about the purpose and use of the stress ball. The stress ball used is made of hygienic, soft silicone material, approximately 6 cm in diameter, and fits in the palm. To avoid negative associations, the tool was referred to as a "squeeze ball." No non-pharmacological interventions will be applied to the control group. In both groups, labor pain will be assessed using the Visual Analog Scale (VAS), and after delivery, the Childbirth Experience Questionnaire (CEQ) will be used to evaluate participants' birth experiences.

Measurement Tools Research data will be collected by face-to-face interview method using Descriptive Information Form, Trauma Follow-up Form, Visual Analogue Scale (VAS) and Birth Experience/Satisfaction Scale (BES).

DETAILED DESCRIPTION:
INTRODUCTION Birth is a natural and unique process that creates significant emotional, social and psychological impacts in women's life cycles. It is emphasized that the pain experienced during this process is universal and is the most severe type of pain a woman can experience. This pain experienced during birth can vary depending on the stages of birth, obstetric care models, psychosocial, environmental, cultural and genetic factors. For this reason, while some women can successfully manage the pain of birth, some women cannot, and they may experience intense stress, lose control over their bodies and feel helpless. However, the World Health Organization (WHO) emphasizes that birth is not only a phenomenon that requires the mother and baby to survive, but also to reach their full potential in terms of health and holistic well-being, and that positive experiences related to birth should be developed.

This study aims to evaluate the effect of stress ball use during the of labor on labor pain and the childbirth experience among primiparous women. The findings obtained may contribute to the literature by demonstrating the effectiveness of stress balls as a non-invasive intervention that can be implemented by nurses and midwives during labor.

MATERIAL AND METHODS Study Design This research is designed as a randomized controlled experimental study. It will be conducted between September and December 2025 with primiparous women admitted to the delivery unit of a public hospital in Turkey.

Population and Sample The study population will consist of primiparous women in the active stage of labor. A simple random sampling method will be used, and 64 primiparous women who meet the inclusion criteria and agree to participate in the study will be included. Participants will be randomly assigned to the intervention group (n=32) or the control group (n=32).

Inclusion Criteria Aged between 18 and 35 years Singleton, viable pregnancy Being primiparous Gestational age between 37 and 42 weeks Having a Visual Analog Scale (VAS) pain score ≥1 during the intrapartum period Absence of systemic or obstetric complications No analgesics or pharmacological pain relief used during labor Exclusion Criteria Having a chronic illness affecting pain perception Difficulty communicating Need for medical intervention during labor (e.g., emergency cesarean section) Ethical Approval and Informed Consent The study will be conducted after receiving approval from the [University/Hospital] Ethics Committee (Approval No: ...). Written permission to use the Childbirth Experience Questionnaire (CEQ) will be obtained from the scale's developer via email. After informing the participants about the study, those who meet the inclusion criteria and agree to participate will be asked to sign an "Informed Consent Form." The research will be carried out in accordance with the principles of the Declaration of Helsinki.

DATA COLLECTION PROCESS Data collection will begin in the latent phase of labor (cervical dilation 1-4 cm). In each phase (active phase, transition phase), participants will be instructed to squeeze the stress ball during contractions accompanied by deep inhalation and to release it during exhalation. During non-contraction periods, their hands will be rested. Participants in the intervention group will be given brief training about the purpose and use of the stress ball. The stress ball used is made of hygienic, soft silicone material, approximately 6 cm in diameter, and fits in the palm. To avoid negative associations, the tool was referred to as a "squeeze ball." No non-pharmacological interventions will be applied to the control group. In both groups, labor pain will be assessed using the Visual Analog Scale (VAS), and after delivery, the Childbirth Experience Questionnaire (CEQ) will be used to evaluate participants' birth experiences.

Measurement Tools

1. Descriptive Information Form; The semi-structured descriptive information form, which was created by the researchers as a result of the literature review, consists of three parts. In the first part, 8 questions determining the sociodemographic characteristics (such as age, education level, family type, language spoken at home, income status, employment status); in the second part, 5 questions determining the characteristics related to pregnancy and childbirth (such as planned pregnancy, regular check-ups during pregnancy, receiving information about normal birth, thoughts and fears); In the third part, there are 5 questions about the non-pharmacological method applied (stress ball application status, being satisfied with the method applied, preferring the method again in subsequent births, experiencing any
2. Visual Analog Scale (VAS) The Visual Analog Scale (VAS) is a simple and widely used tool that allows individuals to subjectively evaluate the intensity of their pain. The scale typically consists of a 10 cm horizontal line, with the left end marked as "no pain" (0) and the right end as "worst possible pain" (10). Participants are asked to indicate their current level of pain by marking a point on the line. This point is then measured with a ruler and converted into a numerical value.

   VAS is considered a reliable and valid instrument for objectively assessing pain perception during labor (Bijur et al., 2001). In this study, pain levels will be measured at specific intervals during the active phase of labor (e.g., at 4 cm, 6 cm, and 8 cm of cervical dilation) using the VAS.
3. Trauma Follow-up Form; This form was developed by the researchers based on the literature review and the Partograph Form (Ghulaxe et al., 2022; Hofmeyr et al., 2021) in order to follow and record the process of the participants from admission to the delivery room until birth. The form includes questions about vaginal examination/touch findings according to the stages of labour, contraction characteristics (start and end times), fetal heart rate, medication status, dose and time of medication used, duration of the second stage of labour, episiotomy and laceration status, Apgar score of the newborn at 1 and 5 minutes, and height-weight status.
4. Childbirth Experience Questionnaire (CEQ)

Development:

The CEQ was developed in Sweden by Dencker and colleagues in 2010. The aim was to create a reliable and valid tool that evaluates women's childbirth experiences in a multidimensional way. The scale was designed to assess the experiences of women who have had vaginal births.

Turkish Adaptation:

Mamuk and colleagues (2019) translated the CEQ into Turkish and conducted validity and reliability studies. With its Turkish adaptation, the scale became usable in childbirth experience research in Turkey.

Structure of the Scale:

The CEQ consists of a total of 22 items and is comprised of four subscales:

Own Capacity Assesses a woman's confidence in her body and herself during childbirth, her ability to cope with labor pain, and her sense of control.

Example item: "I felt that my body was strong during labor." Professional Support Evaluates the quality and adequacy of support provided by healthcare professionals (midwives, nurses, doctors).

Example item: "I was given enough information during labor." Participation Measures the woman's involvement in the childbirth process and whether she was included in decision-making.

Example item: "My opinion was taken into account when decisions were made about the birth." Perceived Safety / Overall Birth Experience Covers the woman's general emotional responses and overall perception of the childbirth process.

Example item: "The birth was a positive experience for me."

Scoring:

The CEQ is structured as a Likert-type scale. Items are scored from 1 to 4:

1. = Strongly disagree
2. = Disagree
3. = Agree
4. = Strongly agree Some items are reverse scored. An average score is calculated for each subscale. Higher scores indicate a more positive childbirth experience.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria

* Aged between 18 and 35 years
* Singleton, viable pregnancy
* Being primiparous
* Gestational age between 37 and 42 weeks
* Having a Visual Analog Scale (VAS) pain score ≥1 during the intrapartum period
* Absence of systemic or obstetric complications
* No analgesics or pharmacological pain relief used during labor

Exclusion Criteria:

* Having a chronic illness affecting pain perception
* Difficulty communicating
* Need for medical intervention during labor (e.g., emergency cesarean section)
* Ethical Approval and Informed Consent
* The study will be conducted after receiving approval from the

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women undergoing labor
Enrollment: 64 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The level of pain experienced during the birth process will be determined with a pain scale consisting of a 10 cc long line divided into equal intervals of 1 cm. It will be checked whether there is a change in the pain scale, which is 10 cm long, | Change in satisfaction with labour pain and labour experience at 12 hours on average during the labour process. Baseline and 12 hours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mamuk, R., Şirin, A., & Kabukçuoğlu, K. (2019). Doğum Deneyim Ölçeği'nin Türkçeye uyarlanması: Geçerlik ve güvenirlik çalışması. Hemşirelikte Eğitim ve Araştırma Dergisi, 16(2), 100-107.
- [Background] Lowe NK. The nature of labor pain. Am J Obstet Gynecol. 2002 May;186(5 Suppl Nature):S16-24. doi: 10.1067/mob.2002.121427. PMID 12011870